CLINICAL TRIAL: NCT04125732
Title: A Phase 1/2 Trial of Direct Administration of AdVEGF-All6A+, a Replication Deficient Adenovirus Vector Expressing a cDNA/Genomic Hybrid of Human VEGF, to the Ischemic Myocardium of Subjects With Angina Pectoris
Brief Title: Epicardial Delivery of XC001 Gene Therapy for Refractory Angina Coronary Treatment (The EXACT Trial)
Acronym: EXACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: XyloCor Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XC001-1001
Record Dates: First submitted 2019-10-04; First posted 2019-10-14 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Ischemia; Angina Refractory; Cardiovascular Diseases; Heart Diseases
Keywords: Refractory angina; Coronary Artery Disease; Gene Therapy
MeSH Terms: conditions — Coronary Artery Disease; Ischemia; Cardiovascular Diseases; Heart Diseases; Angina Pectoris

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AdVEGFXC1 at 1x10^9 vp (Experimental)
  Interventions: Biological: AdVEGFXC1
- AdVEGFXC1 at 1x10^10 vp (Experimental)
  Interventions: Biological: AdVEGFXC1
- AdVEGFXC1 at 4x10^10 vp (Experimental)
  Interventions: Biological: AdVEGFXC1
- AdVEGFXC1 at 1x10^11 vp (Experimental)
  Interventions: Biological: AdVEGFXC1

INTERVENTIONS:
Biological: AdVEGFXC1 — AdVEGFXC1 at one of 4 doses
  Other Names: XC001

SUMMARY:
The primary purpose of this trial is to determine the safety of XC001 (AdVEGFXC1) in patients who suffer from angina caused by coronary artery disease and have no other treatment options. Subjects in this study will receive one of four intramyocardial doses of XC001 that expresses human vascular endothelial growth factor (VEGF) which induces therapeutic angiogenesis (revascularization).

DETAILED DESCRIPTION:
This is a Phase 1/2, first-in-human, multicenter, open-label, single arm dose escalation trial of XC001. Approximately 12 subjects (N=3 per cohort) who have refractory angina will be enrolled into 4 ascending dose groups, followed by an expansion of the highest tolerated dose with 32 additional subjects. XC001 will be administered by a transthoracic epicardial procedure. Safety will be the focus for the initial 6 months after XC001 administration followed by one safety focused telephone evaluation at Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 80 years
* Diagnosis of chronic angina due to obstructive coronary artery disease that is refractory to drug therapy and unsuitable for revascularization via coronary artery bypass graft or percutaneous coronary intervention
* Angina class II-IV based on Canadian Cardiovascular Society Classification of Angina Pectoris
* Adequate hematologic (hemoglobin ≥ 10 g/dL, absolute neutrophil count > 1.2 × 10^3 per μL and platelet count ≥ 75,000 per μL), hepatic (alanine aminotransferase and aspartate aminotransferase ≤ 3 x ULN; total bilirubin ≤ 2 x ULN), and renal function (glomerular filtration rate > 29 mL/minute/1.73 m2)
* Adequate birth control if of child-bearing potential
* Must be willing and able to provide informed consent

Exclusion Criteria:

* ST elevation myocardial infarction (STEMI) or non-ST elevation myocardial infarction (NSTEMI) not requiring revascularization, transmural myocardial infarction or cerebral vascular accident within the past 30 days
* New York Heart Association Function Class III or IV or left ventricular ejection fraction < 25% within the 6 weeks prior to the screening visit
* HbA1c ≥ 8.5%, SBP <90 or >180 mmHg, DBP >100 mmHg
* Other concurrent medical conditions that could jeopardize the safety of the subject or objectives of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint (adverse events) | 6 months
  Safety, as assessed by adverse events and serious adverse events

SECONDARY OUTCOMES:
Secondary Endpoint (Exercise tolerance test) | 6 months
  Exercise tolerance test
Secondary Endpoint (Seattle Angina Questionnaire) | 6 months
  Seattle Angina Questionnaire
Secondary Endpoint (Canadian Cardiovascular Society angina class) | 6 months
  Canadian Cardiovascular Society angina class
Secondary Endpoint (Angina episodes) | 6 months
  Angina episodes

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Stanford University, Stanford, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Cardiology Research Associates, Daytona Beach, Florida
  - University of Florida, Gainesville, Florida
  - James A. Haley VA Medical Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - The Christ Hospital / The Lindner Research Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Houston Methodist, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart DJ, Hilton JD, Arnold JM, Gregoire J, Rivard A, Archer SL, Charbonneau F, Cohen E, Curtis M, Buller CE, Mendelsohn FO, Dib N, Page P, Ducas J, Plante S, Sullivan J, Macko J, Rasmussen C, Kessler PD, Rasmussen HS. Angiogenic gene therapy in patients with nonrevascularizable ischemic heart disease: a phase 2 randomized, controlled trial of AdVEGF(121) (AdVEGF121) versus maximum medical treatment. Gene Ther. 2006 Nov;13(21):1503-11. doi: 10.1038/sj.gt.3302802. Epub 2006 Jun 22. PMID 16791287
- [Derived] Nakamura K, Henry TD, Traverse JH, Latter DA, Mokadam NA, Answini GA, Williams AR, Sun BC, Burke CR, Bakaeen FG, DiCarli MF, Chaitman BR, Peterson MW, Byrnes DG, Ohman EM, Pepine CJ, Crystal RG, Rosengart TK, Kowalewski E, Koch GG, Dittrich HC, Povsic TJ; EXACT Trial Investigators. Angiogenic Gene Therapy for Refractory Angina: Results of the EXACT Phase 2 Trial. Circ Cardiovasc Interv. 2024 May;17(5):e014054. doi: 10.1161/CIRCINTERVENTIONS.124.014054. Epub 2024 May 2. PMID 38696284
- [Derived] Povsic TJ, Henry TD, Traverse JH, Anderson RD, Answini GA, Sun BC, Arnaoutakis GJ, Boudoulas KD, Williams AR, Dittrich HC, Tarka EA, Latter DA, Ohman EM, Peterson MW, Byrnes D, Pepine CJ, DiCarli MF, Crystal RG, Rosengart TK, Mokadam NA. EXACT Trial: Results of the Phase 1 Dose-Escalation Study. Circ Cardiovasc Interv. 2023 Aug;16(8):e012997. doi: 10.1161/CIRCINTERVENTIONS.123.012997. Epub 2023 Jul 28. PMID 37503661
- [Derived] Povsic TJ, Henry TD, Ohman EM, Pepine CJ, Crystal RG, Rosengart TK, Reinhardt RR, Dittrich HC, Traverse JH, Answini GA, Mokadam NA. Epicardial delivery of XC001 gene therapy for refractory angina coronary treatment (The EXACT Trial): Rationale, design, and clinical considerations. Am Heart J. 2021 Nov;241:38-49. doi: 10.1016/j.ahj.2021.06.013. Epub 2021 Jul 2. PMID 34224684